CLINICAL TRIAL: NCT01968070
Title: A Single- and Multiple-Ascending Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of LY3127760 in Healthy Subjects
Brief Title: A Study of LY3127760 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 15181; I7A-MC-EACA (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY3127760; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- LY3127760 (Single) (Experimental): Single oral dose of up to 900 milligram (mg) LY3127760 administered in up to 3 of 3 study periods.
  Interventions: Drug: LY3127760; Drug: Placebo
- Placebo (Single) (Placebo Comparator): Single oral dose of placebo administered in up to 2 of 3 study periods. Placebo matches LY3127760 in appearance.
  Interventions: Drug: LY3127760; Drug: Placebo
- LY3127760 (Multiple) (Experimental): Multiple ascending oral doses of up to 900 mg LY3127760 administered once or twice daily (QD or BID) for 28 days.
  Interventions: Drug: LY3127760; Drug: Placebo
- Placebo (Multiple) (Placebo Comparator): Multiple oral doses of placebo administered QD or BID for 28 days. Placebo matches LY3127760 in appearance.
  Interventions: Drug: LY3127760; Drug: Placebo
- Celecoxib (Multiple) (Active Comparator): Multiple oral doses of 400 mg celecoxib administered QD for 28 days.
  Interventions: Drug: LY3127760; Drug: Celecoxib; Drug: Placebo

INTERVENTIONS:
Drug: LY3127760 — Administered orally
Drug: Celecoxib — Administered orally
  Arms: Celecoxib (Multiple)
Drug: Placebo — Administered orally

SUMMARY:
The main purposes of this study are to evaluate the safety and how well the body handles single and multiple doses of increasing strength of study drug, LY3127760. This study includes three parts. Part 3 may be initiated at sponsor's discretion, based on data from Part 2. Participants will only enroll in 1 of the 3 study parts. This study will last approximately 7 to 13 weeks, depending on part. Screening must be completed within 28 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females as determined by medical history and physical examination
* Male participants agree to use a reliable method of birth control during the study and 3 months following the last dose of the investigational product
* Female participants not of child-bearing potential
* Have a body mass index of 18.5 to 32 kilograms per square meter (kg/m^2) inclusive
* Are normotensive (defined as supine systolic blood pressure [BP] less than 140 millimeters of mercury [mm Hg] and diastolic BP less than 90 mm Hg) without use of any antihypertensives

Exclusion Criteria:

* Have known allergies to LY3127760, related compounds or any components of the formulation, celecoxib or sulfonamides, or history of significant atopy. Participants with known aspirin allergy or allergic reactions to nonsteroidal anti-inflammatory drugs (NSAIDs) should also be excluded
* Have any current or prior history of a significant gastrointestinal illness such as peptic ulcer disease, gastrointestinal (GI) bleeding, chronic gastritis, inflammatory bowel disease or chronic diarrhea
* Have evidence of other chronic liver disease, including but not limited to chronic alcoholic disease, nonalcoholic steatohepatitis, recent history (within 3 months of screening) of acute viral hepatitis or chronic autoimmune hepatitis
* Have used any NSAIDs, celecoxib, aspirin or acetaminophen (at doses greater than 1 gram per day), anticoagulants or antiplatelet agents within 14 days of admission

Part 2 and Part 3 only

* Have 1 plus pretrial pitting edema or 2 plus ankle or pedal edema

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

REFERENCES:
- [Derived] Jin Y, Smith C, Hu L, Coutant DE, Whitehurst K, Phipps K, McNearney TA, Yang X, Ackermann B, Pottanat T, Landschulz W. LY3127760, a Selective Prostaglandin E4 (EP4) Receptor Antagonist, and Celecoxib: A Comparison of Pharmacological Profiles. Clin Transl Sci. 2018 Jan;11(1):46-53. doi: 10.1111/cts.12497. Epub 2017 Aug 30. PMID 28857461

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1 was a single-ascending dose, 2-cohort, 3-period, alternating-group dose-escalation study (cohorts 1-2) and Part 2 of the study was a multiple-ascending dose, 4-cohort, parallel-group, dose-escalation study (cohorts 3-6). Replacement participants received interventions intended for those participants whom discontinued early.
Groups:
- Cohort 1 Sequence 1: Participants received either placebo or 20 milligram (mg) or 200mg LY3127760 capsules orally as per the below dosing sequence.
  Period 1: 20mg LY3127760; Period 2: 200mg LY3127760; Period 3: Placebo;
- Cohort 1 Sequence 2: Participants received either placebo or 20 milligram (mg) or 900mg LY3127760 capsules orally as per the below dosing sequence.
  Period 1: 20mg LY3127760; Period 2: Placebo; Period 3: 900mg LY3127760;
- Cohort 1 Sequence 3: Participants received either placebo or 200 milligram(mg) or 900mg LY3127760 capsules orally as per the below dosing sequence.
  Period 1: Placebo; Period 2: 200 mg LY3127760; Period 3: 900 mg LY3127760;
- Cohort 2 Sequence 1: Participants received either 60mg or 600mg LY3127760 capsules orally as per the below dosing sequence.
  Period 1: 60 mg LY3127760; Period 2: 600 mg LY3127760; Period 3: 600 mg LY3127760 in fasting state;
- Cohort 2 Sequence 2: Participants received either placebo or 60 mg LY3127760 capsules orally as per the below dosing sequence.
  Period 1: 60 mg LY3127760; Period 2: Placebo; Period 3: Placebo;
- Cohort 2 Sequence 3: Participants received either Placebo or 600 mg LY3127760 capsules orally as per the below dosing sequence.
  Period 1: Placebo; Period 2: 600 mg LY3127760; Period 3: 600 mg LY3127760 in fasting state;
- Cohort 3 LY3127760 60mg: Participants received 60mg LY3127760 capsules orally once daily.
- Cohort 3 Placebo; Cohort 4 Placebo; Cohort 5 Placebo; Cohort 6 Placebo: Participants received placebo capsules orally once daily.
- Cohort 3 Celecoxib 400mg; Cohort 4 Celcoxib 400mg; Cohort 5 Celecoxib 400mg; Cohort 6 Celecoxib 400mg: Participants received 400mg Celecoxib capsules orally once daily.
- Cohort 4 LY3127760 200mg: Participants received 200mg LY3127760 capsules orally once daily.
- Cohort 5 LY3127760 20mg: Participants received 20mg LY3127760 capsules orally once daily.
- Cohort 6 LY3127760 600mg: Participants received 300mg LY3127760 capsules orally twice daily.
Period: Period 1
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3 | Cohort 3 LY3127760 60mg | Cohort 3 Placebo | Cohort 3 Celecoxib 400mg | Cohort 4 LY3127760 200mg | Cohort 4 Placebo | Cohort 4 Celcoxib 400mg | Cohort 5 LY3127760 20mg | Cohort 5 Placebo | Cohort 5 Celecoxib 400mg | Cohort 6 LY3127760 600mg | Cohort 6 Placebo | Cohort 6 Celecoxib 400mg
Started | 4 | 4 | 4 | 4 | 4 | 4 | 10 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2
Completed | 4 | 3 | 4 | 2 | 3 | 4 | 8 | 2 | 2 | 9 | 2 | 1 | 9 | 2 | 2 | 8 | 2 | 2
Not Completed | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3 | Cohort 3 LY3127760 60mg | Cohort 3 Placebo | Cohort 3 Celecoxib 400mg | Cohort 4 LY3127760 200mg | Cohort 4 Placebo | Cohort 4 Celcoxib 400mg | Cohort 5 LY3127760 20mg | Cohort 5 Placebo | Cohort 5 Celecoxib 400mg | Cohort 6 LY3127760 600mg | Cohort 6 Placebo | Cohort 6 Celecoxib 400mg
Started | 4 | 4 (1 participant was added to replace the participant who discontinued the period 1.) | 4 | 4 (2 participants were added to replace the 2 participants who discontinued the period 1.) | 3 | 4 | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.) | 0 (Part 2 (Cohorts 3 to 6) was planned only for one period.)
Completed | 4 | 4 | 4 | 4 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3 | Cohort 3 LY3127760 60mg | Cohort 3 Placebo | Cohort 3 Celecoxib 400mg | Cohort 4 LY3127760 200mg | Cohort 4 Placebo | Cohort 4 Celcoxib 400mg | Cohort 5 LY3127760 20mg | Cohort 5 Placebo | Cohort 5 Celecoxib 400mg | Cohort 6 LY3127760 600mg | Cohort 6 Placebo | Cohort 6 Celecoxib 400mg
Started | 4 | 4 | 4 | 4 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 4 | 4 | 4 | 4 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Cohort 6 LY3127760 300mg: Participants received 300mg LY3127760 capsules orally twice daily.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3 | Cohort 3 LY3127760 60mg | Cohort 3 Placebo | Cohort 3 Celecoxib 400mg | Cohort 4 LY3127760 200mg | Cohort 4 Placebo | Cohort 4 Celcoxib 400mg | Cohort 5 LY3127760 20mg | Cohort 5 Placebo | Cohort 5 Celecoxib 400mg | Cohort 6 LY3127760 300mg | Cohort 6 Placebo | Cohort 6 Celecoxib 400mg | Total
Number analyzed (Participants) | 4 | 5 | 4 | 6 | 4 | 4 | 10 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 4 | 6 | 4 | 4 | 10 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 2 | 0 | 4 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 22
  Male | 1 | 3 | 2 | 4 | 2 | 4 | 6 | 1 | 2 | 8 | 2 | 0 | 9 | 1 | 2 | 8 | 1 | 2 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 4 | 6 | 4 | 4 | 10 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 0 | 2 | 1 | 3 | 1 | 1 | 2 | 1 | 1 | 4 | 2 | 1 | 5 | 0 | 1 | 28
  White | 3 | 5 | 1 | 6 | 1 | 2 | 7 | 1 | 1 | 6 | 1 | 1 | 4 | 0 | 1 | 4 | 2 | 1 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 4 | 6 | 4 | 4 | 10 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2 | 9 | 2 | 2 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Data presented are the number of participants who experienced SAEs considered by the investigator to be related to study drug administration. A summary of SAEs and all other non-serious Adverse Event(s) (AEs), regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline to Study Completion (Up To Day 42)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Placebo: Placebo, Single Dose Administered PO
- Part 1: 20 mg LY3127760: 20 mg LY3127760 Single Dose Administered PO
- Part 1: 60 mg LY3127760: 60 mg LY3127760 Single Dose Administered PO
- Part 1: 200 mg LY3127760: 200 mg LY3127760 Single Dose Administered PO
- Part 1: 600 mg LY3127760: 600 mg LY3127760 Single Dose Administered PO
- Part 1: 600 mg LY3127760 (Fasted): 600 mg LY3127760 Single Dose Administered PO During Fasted State
- Part 1: 900 mg LY3127760: 900 mg LY3127760 Single Dose Administered PO
- Part 2: Placebo: Placebo administered PO, once a day (QD), for 28 days.
- Part 2: 20 mg LY3127760: 20 mg LY3127760 administered PO, QD, for 28 days.
- Part 2: 60 mg LY3127760: 60 mg LY3127760 administered PO, QD, for 28 days.
- Part 2: 200 mg LY3127760: 200 mg LY3127760 administered PO, QD, for 28 days.
- Part 2: 300 mg LY3127760: 300 mg LY3127760 administered PO, twice daily (BID), for 28 days.
- Part 2: 400 mg Celecoxib: Celecoxib administered PO, QD, for 28 days.
Arm/Group | Part 1: Placebo | Part 1: 20 mg LY3127760 | Part 1: 60 mg LY3127760 | Part 1: 200 mg LY3127760 | Part 1: 600 mg LY3127760 | Part 1: 600 mg LY3127760 (Fasted) | Part 1: 900 mg LY3127760 | Part 2: Placebo | Part 2: 20 mg LY3127760 | Part 2: 60 mg LY3127760 | Part 2: 200 mg LY3127760 | Part 2: 300 mg LY3127760 | Part 2: 400 mg Celecoxib
Number analyzed (Participants) | 19 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 9 | 10 | 9 | 9 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve Versus Time Curve From Zero to Infinity (AUC 0-∞) of Single Dose LY3127760
Time Frame: Day 1: -1, 0.25, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 96, and 144 Hours
Population: All randomized participants who received at least one dose of study drug for the single dose in Part 1 and had evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms•hour/milliliter (ng•hr/mL)
Groups:
- Part 1: 600 mg LY3127760 (Fasted): 600 mg LY3127760 Single Dose Administered PO During a Fasted State
Arm/Group | Part 1: 20 mg LY3127760 | Part 1: 60 mg LY3127760 | Part 1: 200 mg LY3127760 | Part 1: 600 mg LY3127760 | Part 1: 600 mg LY3127760 (Fasted) | Part 1: 900 mg LY3127760
Number analyzed (Participants) | 8 | 6 | 6 | 8 | 8 | 6
nanograms•hour/milliliter (ng•hr/mL) | NA (NA) — Not calculated because multiple concentrations were below the detection limit of the assay | 3010 (42) | 17200 (9) | 40000 (17) | 47400 (20) | 71900 (20)

3. Secondary Outcome: PK: Maximum Observed Concentration (Cmax) of Single Dose LY3127760
Time Frame: Day 1: -1, 0.25, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 96, and 144 Hours
Population: All randomized participants who received at least one dose of study drug for the single dose in Part 1 and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Part 1: 20 mg LY3127760 | Part 1: 60 mg LY3127760 | Part 1: 200 mg LY3127760 | Part 1: 600 mg LY3127760 | Part 1: 600 mg LY3127760 (Fasted) | Part 1: 900 mg LY3127760
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
nanograms/milliliter (ng/mL) | 264 (41) | 890 (19) | 3880 (33) | 10300 (37) | 18900 (40) | 21600 (27)

4. Secondary Outcome: PK: Time of Maximum Observed Concentration (Tmax) of Single Dose LY3127760
Time Frame: Day 1: -1, 0.25, 0.5, 1, 2, 4, 8, 12, 16, 24, 36, 48, 96, and 144 Hours
Population: All randomized participants who received at least one dose of study drug for the single dose in Part 1 and had evaluable Tmax data.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1: 20 mg LY3127760 | Part 1: 60 mg LY3127760 | Part 1: 200 mg LY3127760 | Part 1: 600 mg LY3127760 | Part 1: 600 mg LY3127760 (Fasted) | Part 1: 900 mg LY3127760
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Hour | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.02] | 2.00 [0.25 to 4.00] | 2.00 [2.00 to 4.00] | 1.00 [0.52 to 2.00] | 1.50 [1.00 to 2.00]

5. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve During One Dosing Interval [AUC-tau (τ)] of Multiple Doses LY3127760
Description: AUC-tau (τ) where τ is 24-hours for the 20 mg, 60 mg, and 200 mg cohorts, and 12-hours for the 300 mg cohort.
Time Frame: Day 28: -1, 0.25, 0.5, 1, 2, 4, 8, 12, 16, and 24 Hours
Population: All randomized participants who received at least one dose of study drug for multiple dosing in Part 2 and had evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/ml
Groups:
- Part 2: 20 mg LY3127760: 20 mg LY3127760 Administered QD PO, Day 1-28
- Part 2: 60 mg LY3127760: 60 mg LY3127760 Administered QD PO, Day 1-28
- Part 2: 200 mg LY3127760: 200 mg LY3127760 Administered QD PO, Day 1-28
- Part 2: 300 mg LY3127760: 300 mg LY3127760 Administered BID PO, Day 1-28
Arm/Group | Part 2: 20 mg LY3127760 | Part 2: 60 mg LY3127760 | Part 2: 200 mg LY3127760 | Part 2: 300 mg LY3127760
Number analyzed (Participants) | 9 | 8 | 9 | 8
ng•hr/ml | 1020 (20) | 4350 (50) | 11300 (23) | 19700 (15)

6. Secondary Outcome: PK: Cmax of Multiple Doses LY3127760
Time Frame: Post last dose on Day 28: 0.25, 0.5, 1, 2, 4, 8, 12, 16, 24, 72, and 168 Hours
Population: All randomized participants who received at least one dose of study drug for multiple dosing in Part 2 and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: 20 mg LY3127760 | Part 2: 60 mg LY3127760 | Part 2: 200 mg LY3127760 | Part 2: 300 mg LY3127760
Number analyzed (Participants) | 9 | 8 | 9 | 8
ng/mL | 301 (19) | 1210 (53) | 3650 (27) | 6170 (22)

7. Secondary Outcome: PK: Tmax of Multiple Doses LY3127760
Time Frame: Post-last dose on Day 28: 0.25, 0.5, 1, 2, 4, 8, 12, 16, 24, 72, and 168 Hours
Population: All randomized participants who received at least one dose of study drug for multiple dosing in Part 2 and had evaluable Tmax data.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 2: 20 mg LY3127760 | Part 2: 60 mg LY3127760 | Part 2: 200 mg LY3127760 | Part 2: 300 mg LY3127760
Number analyzed (Participants) | 9 | 8 | 9 | 8
hour | 2.00 [1.00 to 4.00] | 1.65 [1.00 to 4.00] | 2.00 [1.00 to 2.02] | 2.00 [1.00 to 2.00]

ADVERSE EVENTS:
Description: Two participants were randomized into a Part 1 scheme where they received placebo 2 out of the 3 dosing periods. Those participants are represented only once in the placebo arm in adverse events.
Groups:
- Placebo (Part 1): Placebo, Single Dose Administered PO
- 20 mg LY3127760 (Part 1): 20 mg LY3127760 Single Dose Administered PO
- 60 mg LY3127760 (Part 1): 60 mg LY3127760 Single Dose Administered PO
- 200 mg LY3127760 (Part 1): 200 mg LY3127760 Single Dose Administered PO
- 600 mg LY3127760 (Part 1): 600 mg LY3127760 Single Dose Administered PO
- 600 mg LY3127760 (Fasted) (Part 1): 600 mg LY3127760 Single Dose Administered PO During Fasted State
- 900 mg LY3127760 (Part 1): 900 mg LY3127760 Single Dose Administered PO
- Placebo (Part 2): Placebo, Administered QD PO, Day 1-28
- 20 mg LY3127760 (Part 2): 20 mg LY3127760 Administered QD PO, Day 1-28
- 60 mg LY3127760 (Part 2): 60 mg LY3127760 Administered QD PO, Day 1-28
- 200 mg LY3127760 (Part 2): 200 mg LY3127760 Administered QD PO, Day 1-28
- 300 mg LY3127760 (Part 2): 300 mg LY3127760 Administered BID PO, Day 1-28
- 400 mg Celecoxib (Part 2): 400 mg celecoxib Administered QD PO, Day 1-28
Arm/Group | Placebo (Part 1) | 20 mg LY3127760 (Part 1) | 60 mg LY3127760 (Part 1) | 200 mg LY3127760 (Part 1) | 600 mg LY3127760 (Part 1) | 600 mg LY3127760 (Fasted) (Part 1) | 900 mg LY3127760 (Part 1) | Placebo (Part 2) | 20 mg LY3127760 (Part 2) | 60 mg LY3127760 (Part 2) | 200 mg LY3127760 (Part 2) | 300 mg LY3127760 (Part 2) | 400 mg Celecoxib (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/9 | 0/10 | 0/9 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 4/19 | 2/8 | 1/8 | 1/8 | 3/8 | 1/8 | 2/8 | 2/8 | 4/9 | 5/10 | 4/9 | 6/9 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part 1) (N=19) | 20 mg LY3127760 (Part 1) (N=8) | 60 mg LY3127760 (Part 1) (N=8) | 200 mg LY3127760 (Part 1) (N=8) | 600 mg LY3127760 (Part 1) (N=8) | 600 mg LY3127760 (Fasted) (Part 1) (N=8) | 900 mg LY3127760 (Part 1) (N=8) | Placebo (Part 2) (N=8) | 20 mg LY3127760 (Part 2) (N=9) | 60 mg LY3127760 (Part 2) (N=10) | 200 mg LY3127760 (Part 2) (N=9) | 300 mg LY3127760 (Part 2) (N=9) | 400 mg Celecoxib (Part 2) (N=8)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days